CLINICAL TRIAL: NCT03920423
Title: Impact Factors to Success Without Posterior Wall Puncture Using Ultrasound-guided Short-axis Out-of-plane Dynamic Approach
Brief Title: Impact Factors to Success Without Posterior Wall Puncture Using Dynamic Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1338
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Radial Artery Catheterization; Ultrasound or Ultrasonography; Ultrasound-guided Short-axis Out-of-plane Dynamic Approach

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shallow depth (No Intervention): Radial arterial deth is shallow than the cutoff point that relative to results.
- improved depth (Experimental): Radial arterial deth is shallow than the cutoff point that relative to results, and increased by injection of saline to more than deep cutoff point.
  Interventions: Procedure: improvement of arterial depth

INTERVENTIONS:
Procedure: improvement of arterial depth — deepen radial arterial depth by injection of saline to more than deep cutoff point relative to result.
  Arms: improved depth

SUMMARY:
The study is designed to evaluate and validate impact factors to success and complication using ultrasound guided short-axis out-of-plane dynamic approach, and validate the impaction.

DETAILED DESCRIPTION:
The study including two phase: observational phase and validation phase. In observational phase, factors relative to success catheterization without posterior puncture and success in first attempt are evaluated. In validation phase, patients are randomized into different depth group with or without injection of saline. Success without posterior wall puncture, success in first attempt and overall, catheterization time are compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* requirement of radial arterial catheterization during perioperative period
* within cardiac-vascular disease
* written consent

Exclusion Criteria:

* contraindication to radial arterial catheterization
* abnormal artery evaluated by ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
success without posterior wall puncture | Through study completion,an average of 5 minutes
  success to puncture and catheterize of radial artery, without posterior wall puncture.
success in first attempt | Through study completion,an average of 5 minutes
  success puncture and catheterization in first attempt

SECONDARY OUTCOMES:
success overall | Through study completion,an average of 5 minutes
  success catheterization with the maximum of 10 minutes
time needed to catheterization | Through study completion,an average of 5 minutes
  time required for successful puncturing and catheterization with the maximum of 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No